CLINICAL TRIAL: NCT06071806
Title: The Application of Topical 5-Fluorouracil to Reduce the Recurrence of Odontogenic Keratocyst
Brief Title: Recurrence of Odontogenic Keratocyst
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed Kamal Eid Allam, Associate professor, Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R-OS-12-22-2
Record Dates: First submitted 2023-09-24; First posted 2023-10-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Odontogenic Cyst
Keywords: Odontogenic Keratocyst; 5- Fluorouracil; Recurrence
MeSH Terms: conditions — Odontogenic Cysts; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- surgery/Topical application of fluorouracil (Other): The entire cyst lining radically enucleated with peripheral ostectomy was carried out for all bony walls to remove the microscopic satellite cyst, a sterile radiopaque quarter-inch ribbon gauze coated with 5-FU cream was packed into the surgical wound. Closure of the wound was then done in the usual manner using 3/0 vicryl leaving approximately1 cm of a small distal end of the gauze exposed to allow for easy removal after 24 hours postoperatively
  Interventions: Other: Topical Application of 5-Fluorouracil

INTERVENTIONS:
Other: Topical Application of 5-Fluorouracil — The entire cyst lining radically enucleated in conjunction with any overlying mucosa, followed by extensive cavity thorough curettage, peripheral ostectomy was carried out for all bony walls to remove the microscopic satellite cyst, with identification, isolation, retraction, and preservation of the lingual and inferior alveolar bundle,a sterile radiopaque quarter-inch ribbon gauze coated with 5-FU cream was packed into the surgical wound. Closure of the wound was then done in the usual manner using 3/0 vicryl leaving approximately1 cm of a small distal end of the gauze exposed to allow for easy removal after 24 hours postoperatively

SUMMARY:
The aim of current cross over clinical trial is to evaluate the effect of topical 5-FU as adjunct therapy in reducing risk of the recurrence of OKCs

DETAILED DESCRIPTION:
The main inclusion criteria in this study will be 48 patients with biopsy proved odontogenic keratocyst with no relevant systemic diseases which might affect healing process. patients will be treated with 5-FU cream (Efudex; Valeant Inc, Laval, Quebec, Canada) after enucleation and peripheral ostectomy of the odontogenic keratocyst.

* A detailed preoperative assessment for all patients will be carried out including history taking, clinical and radiographical examination.
* All surgical procedures will be carried out under general anesthesia with nasal endotracheal intubation.
* Through an intraoral incision, the full thickness mucoperiosteal flap will be raised. The entire cyst lining radically enucleated in conjunction with any overlying mucosa, followed by extensive cavity thorough curettage with meticulous evaluation of any residual daughter cyst lining with reduction of the lingual and buccal undercut bony walls to remove residual macroscopic cystic epithelium.
* After enucleation and peripheral ostectomy of the OKC lesion, a sterile radiopaque quarter-inch ribbon gauze is coated with 5-FU cream and packed into the surgical wound. The wound is closed in the usual manner using 3/0 vicryl leaving a small distal end (approximately1 cm) of gauze exposed to allow for gauze removal at 24 hours postoperatively.

All patients will be regularly followed up for 12 months postoperatively clinically and radiographically

ELIGIBILITY:
Inclusion Criteria:

* patients with biopsy proved odontogenic keratocyst

Exclusion Criteria:

* relevant systemic diseases which might affect healing process.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2022-12-02 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
degree of pain | 6 month
  pain is measured on a visual analogue scale (VAS) started from 0 which represent (no pain at all) and end by 10 which represent (most severe pain)
swelling | 6 month
  Swelling is assessed using a vertical and horizontal references with a tape on four reference points; outer canthus of the eye, angle of the mandible, tragus, and outer corner of the mouth

SECONDARY OUTCOMES:
Quantitative computed tomography (CT) | 12 month
  Quantitative interpretation of values derived from Hounsfield units with a suitable calibration procedure is the modality of choice to determine the local bone mineral density during the follow up periods

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed K Allam, Ass prof, Principal Investigator — Tanta University
Locations (1):
- Tanta University, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No